CLINICAL TRIAL: NCT01808027
Title: Evaluation of the Methods and Management of Acute Coronary Events: 3. Investigating Variation in Hospital Acute Coronary Syndrome Outcomes
Brief Title: Investigating Variation in Hospital Acute Coronary Syndrome Outcomes
Status: Completed | Type: Observational
Sponsor: University of Leeds (Other)
Responsible Party: Principal Investigator, Oras Alabas, Dr, University of Leeds
Other Study IDs: 10/H1313/74
Record Dates: First submitted 2013-03-07; First posted 2013-03-08 (Estimated); Last update posted 2013-03-08 (Estimated); Status verified 2013-03

CONDITIONS: Acute Myocardial Infarction
Keywords: quality of life drug adherence drug compliance mortality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Acute myocardial infarction: patient with suspected acute coronary syndrome (ACS).

SUMMARY:
To investigate the causes of hospital variation in outcomes from acute coronary syndromes in England and develop recommendations for improving patient care.

DETAILED DESCRIPTION:
Over the last few years the chance of dying from a heart attack in England and Wales has reduced dramatically. Even so, there remain huge differences in mortality between hospitals. For example, up to a third of patients with a heart attack who attend hospitals in England are more likely to die than would be expected. That is, the type of treatment and the risk of death depends upon where a patient lives and which hospital they attend. In part, the variation in death may be due to the services available at the hospital or to factors such as socioeconomic deprivation. It may also relate to other factors such as depression, cardiac rehabilitation and whether patients take their medication after discharge from hospital. Using powerful statistical approaches that include measures of quality of life, we propose to examine data about heart attacks in England and investigate the 'postcode lottery of care'. Our aim, using regional data about heart attacks is to identify and measure the effects of hospital care. This research will identify hospital qualities that promote improved patient care. In doing so, best practice will be highlighted and healthcare policy changed so that all patients will have an equal chance of surviving a heart attack.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Both sexes
* Acute admission to the acute Trust with suspected acute coronary syndrome

Exclusion Criteria:

* Patients at a terminal stage of any illness
* Those in whom follow up would be inappropriate or impractical

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consented patients with acute coronary syndrome were recruited from acute Trusts in England. These hospitals have been selected because of their diverse population demographics, different acute coronary syndrome care pathways and established track record for good data collection. Specifically these hospitals represent both teaching hospitals and community hospitals - but more importantly include a wide range of patient types. Mortality tracked through the UK statistics authority, and primary and secondary endpoints tracked locally and transferred through the secure NHS net to a central database.
Sampling Method: Non-Probability Sample
Enrollment: 5555 (Actual)
Dates: Start 2011-02; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
delays to treatment | 12 months
  Quantification of hospital attributable effects relating to early and late mortality

SECONDARY OUTCOMES:
Describing trajectories of quality of life recovery patterns | 12 month
  Describing trajectories of quality of life recovery patterns

OTHER OUTCOMES:
Develop a risk score and a near-point risk Acute Coronary Syndrome model | two years
  Develop a risk score and a near-point risk Acute Coronary Syndrome model

CONTACTS AND LOCATIONS:
Overall Officials: Chris P Gale, PhD, Principal Investigator — University of Leeds
Locations (1):
- University of Leeds, Leeds, West Yorkshire, United Kingdom

REFERENCES:
- [Derived] Munyombwe T, Dondo TB, Hall M, Nadarajah R, Hurdus B, Aktaa S, Haris M, Keeley A, West R, Hall A, Norman P, Gale CP. Cohort profile: Evaluation of the Methods and Management of Acute Coronary Events (EMMACE) Longitudinal Cohort. Eur Heart J Qual Care Clin Outcomes. 2023 Aug 7;9(5):442-446. doi: 10.1093/ehjqcco/qcad040. PMID 37451698
- [Derived] Dondo TB, Munyombwe T, Hall M, Hurdus B, Soloveva A, Oliver G, Aktaa S, West RM, Hall AS, Gale CP. Sex differences in health-related quality of life trajectories following myocardial infarction: national longitudinal cohort study. BMJ Open. 2022 Nov 8;12(11):e062508. doi: 10.1136/bmjopen-2022-062508. PMID 36351712
- [Derived] Munyombwe T, Dondo TB, Aktaa S, Wilkinson C, Hall M, Hurdus B, Oliver G, West RM, Hall AS, Gale CP. Association of multimorbidity and changes in health-related quality of life following myocardial infarction: a UK multicentre longitudinal patient-reported outcomes study. BMC Med. 2021 Sep 28;19(1):227. doi: 10.1186/s12916-021-02098-y. PMID 34579718
- [Derived] Hurdus B, Munyombwe T, Dondo TB, Aktaa S, Oliver G, Hall M, Doherty P, Hall AS, Gale CP. Association of cardiac rehabilitation and health-related quality of life following acute myocardial infarction. Heart. 2020 Nov;106(22):1726-1731. doi: 10.1136/heartjnl-2020-316920. Epub 2020 Aug 21. PMID 32826289
- [Derived] Munyombwe T, Hall M, Dondo TB, Alabas OA, Gerard O, West RM, Pujades-Rodriguez M, Hall A, Gale CP. Quality of life trajectories in survivors of acute myocardial infarction: a national longitudinal study. Heart. 2020 Jan;106(1):33-39. doi: 10.1136/heartjnl-2019-315510. Epub 2019 Nov 7. PMID 31699696
- [Derived] Alabas OA, West RM, Gillott RG, Khatib R, Hall AS, Gale CP; EMMACE-3 Investigators. Evaluation of the Methods and Management of Acute Coronary Events (EMMACE)-3: protocol for a longitudinal study. BMJ Open. 2015 Jun 23;5(6):e006256. doi: 10.1136/bmjopen-2014-006256. PMID 26105029